CLINICAL TRIAL: NCT04187352
Title: A Multi-Center, Double-Blind, Randomized, Phase III Study to Investigate the Efficacy and Safety of CS1001 in Combination With Fluorouracil and Cisplatin (FP) Compared to Placebo in Combination With FP as First-Line Therapy in Subjects With Unresectable Locally Advanced, Recurrent or Metastatic Esophageal Squamous Cell Carcinoma (ESCC)
Brief Title: A Study of CS1001 in Subjects With Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS1001-304
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Unresectable Locally Advanced, Recurrent or Metastatic Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Recurrence; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CS1001+ Fluorouracil+Cisplatin (Experimental)
  Interventions: Drug: CS1001+ Fluorouracil+Cisplatin
- Placebo+ Fluorouracil+Cisplatin (Active Comparator)
  Interventions: Drug: Placebo+ Fluorouracil+Cisplatin

INTERVENTIONS:
Drug: CS1001+ Fluorouracil+Cisplatin — CS1001 1200 mg, intravenous infusion on the first day of each cycle (3 weeks) (Q3W).
  Fluorouracil: 800 mg/m2/day, continuous intravenous infusion on Day 1 to Day 4 of each cycle Cisplatin: 80 mg/m2, intravenous infusion on the first day of each cycle.
  Arms: CS1001+ Fluorouracil+Cisplatin
Drug: Placebo+ Fluorouracil+Cisplatin — Placebo 1200 mg, intravenous infusion on the first day of each cycle (3 weeks) (Q3W).
  Fluorouracil: 800 mg/m2/day, continuous intravenous infusion on Day 1 to Day 4 of each cycle Cisplatin: 80 mg/m2, intravenous infusion on the first day of each cycle.
  Arms: Placebo+ Fluorouracil+Cisplatin

SUMMARY:
Phase III Study to Investigate the Efficacy and Safety of CS1001 or Placebo in Combination with FP as First-Line Therapy in Subjects with Unresectable Locally Advanced, Recurrent or Metastatic Esophageal Squamous Cell Carcinoma

ELIGIBILITY:
Inclusion criteria

1. ≥ 18 years and ≤ 75 years on the day of signing informed consent form (ICF).
2. Fully informed of the study, with good compliance and willing to provide written ICF. The ICF must be signed before performing any protocol-related procedure (that is not a part of subject's routine medical care).
3. Subjects with pathohistologically or cytologically confirmed unresectable locally advanced, relapsed or metastatic ESCC (based on American Joint Committee on Cancer [AJCC] Guideline version 8, see Appendix 14.2)
4. Subjects must not be eligible for radical therapy such as radical chemoradiotherapy or surgery.
5. Subjects who have not received any systemic anti-neoplastic therapy as the main regimen for locally advanced or metastatic ESCC. (Subjects who received prior neoadjuvant, adjuvant or radical chemoradiotherapy for ESCC but had relapse or progression of disease 6 months after the completion of these treatments are allowed.)
6. ECOG PS 0 or 1.
7. Life expectancy ≥ 3 months.
8. Subjects have at least one measurable lesion as evaluated by the investigator according to RECIST v1.1, and the baseline imaging assessment must be performed within 28 days prior to the first dose of investigational product. Target lesions in the past radiation fields, if confirmed as radiological progression, are considered as measurable lesions.
9. Palliative treatment (e.g. radiotherapy) for local lesion must be completed ≥ 14 days prior to the first dose of investigational product.
10. Subjects must provide tumor tissue samples (formalin fixed-paraffin embedded [FFPE] tissue block or unstained tumor tissue sections) for biomarker analysis, in order to determine the expression of PD-L1.
11. Subjects must have adequate organ function as assessed in the following laboratory tests (subjects must not receive any blood transfusion or any hematopoietic growth factor within 7 days prior to the test)
12. Female subjects with childbearing potential (unless with documentation of sterilization surgery or being post-menopausal) must have negative serum pregnancy test result at screening. Female subject with childbearing potential (unless with documentation of sterilization surgery or being post-menopausal) or male subjects and their partners must agree to use an effective contraceptive measure from the day of signing ICF till at least 6 months after the last dose of investigational product.

Exclusion criteria

1. Adenocarcinoma, mixture of adenocarcinoma and squamous cell carcinoma, or other pathological type of esophageal cancer.
2. Subjects with active central nervous system (CNS) metastasis and/or carcinomatous meningitis (that is symptomatic, or requires treatment, or no radiological evidence confirming the stability of the lesion within 28 days prior to the first dose of investigational product).
3. With another active primary malignancy in the past 5 years, except local curable cancers that have undergone curative therapy, e.g. basal cell carcinoma of skin, squamous cell carcinoma of skin, superficial bladder cancer, prostate cancer in situ, breast cancer in situ or cervical cancer in situ.
4. Known history of positive human immunodeficiency virus (HIV) test result or acquired immunodeficiency syndrome (AIDS).
5. Any severe or uncontrolled systemic disease, e.g., diabetes mellitus or hypertension, that may increase the risk associated with participation in the study or investigational product administration, or compromise subject's ability to receive investigational product, as per investigator's judgment.
6. Subjects who have previously received any treatment of antibody or drug that targets at T-cell coregulatory pathways or immune checkpoint pathways, e.g., antibodies targeting at programmed death receptor-1 (PD-1), programmed death receptor-ligand 1 (PD-L1), cytotoxic T lymphocyte-associated antigen 4 (CTLA-4), OX-40, CD137, T cell immunoglobulin mucin molecule 3 (TIM-3), lymphocyte activation gene 3 (LAG-3), etc. Subjects who have received cell-based immunotherapy (e.g., cytokine-induced killer cell [CIK], chimeric antigen receptor T cell [CAR-T] immunotherapy, etc.).
7. All toxicities except for alopecia and fatigue that are caused by the prior anti-neoplastic treatment has recovered to Grade 1 (according to National Cancer Institute Common Toxicity Criteria for Adverse Events [NCI CTCAE] v5.0).
8. Subjects with history of allogenic stem cell or solid organ transplantation.
9. Subjects with any condition that in the investigator's opinion are not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by Blinded Independent Central Review (BICR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Approximately 43 months from the time of randomization
  PFS was defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 as assessed by BICR, or death due to any cause, whichever occurred first.
Overall survival (OS) | Approximately 43 months from the time of randomization
  OS was defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
PFS assessed by investigators according to RECIST v1.1 | Approximately 43 months from the time of randomization
  PFS was defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 as assessed by investigators, or death due to any cause, whichever occurred first.
Objective response rate (ORR) assessed by BICR and investigators according to RECIST v1.1 | Approximately 43 months from the time of randomization
  ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR) or a Partial Response (PR) per RECIST 1.1.
Duration of response (DoR) assessed by BICR and investigators according to RECIST v1.1 | Approximately 43 months from the time of randomization
  DOR was defined as the time from first documented evidence of confirmed CR or PR until PD or death due to any cause, whichever occurred first.

CONTACTS AND LOCATIONS:
Locations (72):
- China (72):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Hefei Second People's Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Peaking University International Hospital, Beijing, Beijing Municipality
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - Special Medical Center of The People's Liberation Army of China, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Jieyang People's Hospital, Jieyang, Guangdong
  - Affiliated Tumor Hospital of Shantou University Medical College, Shantou, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat sen University, Zhuhai, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - Handan Central Hospital, Handan, Hebei
  - Shijiazhuang People's Hospital, Shijiazhuang, Hebei
  - The Affiliated Tumor Hospital of Harbin Meidical University, Haerbin, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - Nanyang First People's Hospital, Nanyang, Henan
  - Puyang Oilfield General Hospital, Puyang, Henan
  - Xinxiang First People's Hospital, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Tongji Medical College of HUST, Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Fifth Hospital, Wuhan, Hubei
  - Wuhan Union Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Changzhou Tumor Hospital, Changzhou, Jiangsu
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Tonghua Central Hospital, Tonghua, Jilin
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Jinan central Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Linfen Central Hospital, Linfen, Shanxi
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Chengdu Fifith people's hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Yibin Second People's Hospital, Yibin, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Cancer Hospital Affiliated to Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Li J, Chen Z, Bai Y, Liu B, Li Q, Zhang J, Zhou J, Deng T, Zhou F, Gao S, Yang S, Ye F, Chen L, Bai W, Yin X, Cang S, Liu L, Pan Y, Luo H, Ji Y, Zhang Z, Wang J, Yang Q, Li N, Huang R, Qu C, Ni J, Wang B, Xu Y, Hu J, Shi Q, Yang J. First-line sugemalimab with chemotherapy for advanced esophageal squamous cell carcinoma: a randomized phase 3 study. Nat Med. 2024 Mar;30(3):740-748. doi: 10.1038/s41591-024-02797-y. Epub 2024 Feb 1. PMID 38302715